CLINICAL TRIAL: NCT03798288
Title: A Decision Support System for Self-management of Low Back Pain - a Randomized Controlled Trial for the selfBACK Project
Brief Title: Randomised Controlled Trial for the selfBACK Project
Acronym: selfBACK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Norwegian University of Science and Technology (Other); National Research Centre for the Working Environment, Denmark (Other Government); University of Glasgow (Other); Robert Gordon University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18/17955CDJ
Record Dates: First submitted 2019-01-07; First posted 2019-01-09 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Low Back Pain
Keywords: Digital Decision Support System; App; Self-management
MeSH Terms: conditions — Low Back Pain; Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: The study design is a multi-center randomised controlled trial with 2 parallel arms
Who Masked: Investigator
Masking Description: The analysis of the data will be performed blindly.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care + selfBACK (Experimental): The selfBACK system constitutes a data-driven decision support system that uses case-based reasoning to capture and reuse participant cases to suggest the most suitable self-management plan for participants. The system is an intelligent system delivering self-management plans tailored to individual participant characteristics. Information about participant characteristics is collected via a (baseline) questionnaire, weekly self-reports via the app on symptom progression etc., and a wristband that detect daily number of steps. The weekly plans are presented in an app to participants.
  The weekly plan includes three categories of content;
  1. information/education
  2. recommended daily number of steps
  3. recommended strength and flexibility exercises
  Interventions: Behavioral: selfBACK; Other: Usual care
- Usual care (Active Comparator): Any diagnostic or treatment-related pathway (e.g. receive information, advice or treatment) as instructed by their health care professional. Patients are allowed to seek care, treatment or help elsewhere as normal.
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: selfBACK — Participants will use the selfBACK system and app in addition to receiving usual care
  Arms: Usual care + selfBACK
Other: Usual care — Participants will receive usual care

SUMMARY:
The intervention consists of a digital decision support system delivering a weekly plan of suggested activities that the participant can use to self-manage their low back pain (LBP) via an smartphone app.

DETAILED DESCRIPTION:
The selfBACK intervention consists of the selfBACK system, that provides the participants with an individually tailored weekly plan of suggested activities to use in their self-management of low back pain.

The selfBACK system constitutes a data-driven decision support system that uses case-based reasoning to capture and reuse participant cases to suggest the most suitable self-management plan for participants. The system is an intelligent system delivering self-management plans tailored to individual participant characteristics. Information about participant characteristics is collected via a (baseline) questionnaire, weekly self-reports via the app on symptom progression etc., and a wristband that detect daily number of steps. The weekly plans are presented in an app to participants.

The weekly plan includes three categories of content;

1. information/education
2. recommended daily number of steps
3. recommended strength and flexibility exercises

Outcomes are collected as baseline, 6 weeks, 3, 6, 9 months.

ELIGIBILITY:
Inclusion Criteria:

* Seeking care from primary health-care practice (general practitioners, physiotherapists, chiropractors) or a local outpatient spinecenter (DK) for non-specific LBP within the past 8 weeks
* LBP of any duration
* Mild-to severe pain-related disability rated as 6 or above on the Roland Morris Disability Questionnaire
* Age: ≥18 years
* Own and regularly use a smart phone (with at least Android 7.0 or iOS11.0) with internet access (Wi-Fi and/or mobile data)
* Have a working email address and have access to a computer with internet access to complete questionnaires in a web browser.

Exclusion Criteria:

* Not interested,
* Unable to speak, read or understand the national language (Danish/ Norwegian),
* Cognitive impairments or learning disabilities limiting participation,
* Mental or physical illness or condition limiting participation,
* Inability to take part in exercise/physical activity,
* Fibromyalgia (diagnosed by a health care professional),
* Pregnancy,
* Previous back surgery
* Ongoing participation in other research trials for LBP management.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 461 (Actual)
Dates: Start 2019-03-08 (Actual); Primary Completion 2020-05-06 (Actual); Study Completion 2020-10-20 (Actual)

PRIMARY OUTCOMES:
Roland Morris Disability Questionnaire | change from baseline to 3 months
  The primary outcome is the Roland Morris Disability Questionnaire (RMDQ) assessing pain-related disability. The questionnaire includes 24 items asking participants to indicate if they experience functional impairments by answering "yes" or "no" to a series of descriptions of functional abilities with higher scores indicating higher level of disability.

SECONDARY OUTCOMES:
Pain Self-Efficacy Questionnaire | change from baseline to 3 months
  The questionnaire assesses the participant's level of confidence in carrying out specific activities despite their pain. The PSEQ is a 10-item questionnaire scored on an ordinal scale ranging from zero [completely disagree] to six [completely agree].
The Fear Avoidance Belief Questionnaire | change from baseline to 3 months
  The FABQ is a 5-item questionnaire, where the participants score their beliefs about their LBP on an ordinal scale ranging from zero [completely disagree] to six [completely agree]
Pain intensity | change from baseline to 3 months
  Pain intensity measured as average and worst LBP within the past week. Measured on a 0 - 10 Numerical Rating Scale with 0 being no pain and 10 being worst pain imaginable.
Brief Illness Perception Questionnaire | change from baseline to 3 months
  The questionnaire evaluates the participants' illness perception in an 8-item questionnaire. Items are scored on an ordinal scale ranging from zero [no problems] to 10 [worst severity].
Saltin-Grimby Physical Activity Level Scale | change from baseline to 3 months
  Participants indicate their amount of time per week performing leisure activities with four levels of intensity ranging from sedentary to vigorous physically active
Patients Global Perceived Effect | 3 months
  A single item question for Patient's Global Perceived Effect will be asked at follow-up, where participants are asked to rate improvement or deterioration of their LBP compared to before the intervention

OTHER OUTCOMES:
Workability | change from baseline to 3 months
  Workability is measured by a single-item and rated on an 11-point NRS scale ranging from zero [completely unable to work] to 10 [work ability at its best].
Health-related Quality of Life | change from baseline to 3 months
  The EuroQoL 5-dimension (EQ-5D) questionnaire is used to asses quality of life within each of the five dimension (i.e., mobility, self-care, activities, pain/discomfort and anxiety/depression).
Activity limitation | change from baseline to 3 months
  Activity Limitation evaluates if LBP has limited work and leisure time activities. The questionnaire consists of two single items with response options "yes" and "no".
Sleep | change from baseline to 3 months
  Sleep is assessed by self-report using four items concerning problems with falling asleep, waking up repeatedly, waking up too early, and feeling sleepy during the day.
Perceived Stress Scale | change from baseline to 3 months
  a 10-item questionnaire asking about frequency of thoughts and feelings related to perceived stress
Patient Health Questionnaire-8 | change from baseline to 3 months
  the questionnaire is an 8-item questionnaire used to evaluate the participants' depressive symptoms. Items are scored on a 4-point Likert scale scoring frequency of experiencing symptoms of depression.
Patient Specific Functional Scale | change from baseline to 3 months
  Participants rate their function on up to two self-selected activities, are asked to rate if they are unable to do or are having difficulty with the their ability to perform self-selected activities regarded as important by the participants themselves
Pain duration and frequency | change from baseline to 3 months
  Pain duration measures patients' self-reported length of current pain episode. Pain medication measures the frequency of the non-prescription pain medication use for LBP.
Virtual Care Climate Questionnaire | 4 months
  The Virtual Care Climate Questionnaire concerns patients' perceived support for autonomy in a virtual care setting.
User ratings | 4 months
  Three rating questions on overall rating, ease of use and recommendation to others scored on a 5-point system
Tailoring variables | weekly for 9 months
  Participants in the intervention are on a weekly basis asked a set of tailoring questions. These are tracked over the intervention period. The tailoring questions include items on lob back pain (NRS for pain intensity), function, fear-avoidance, workability, sleep, pain self-efficacy, stress, symptoms of depression, and barriers for self-management.
  Note. not all questions are asked on a weekly basis
Physical activity | weekly for 9 months
  The patients' weekly recommended step count goal, and the actual achieved step count per. day
Exercise volume | weekly for 9 months
  The patients report back their completed exercise volume as number of sets and repetitions for their suggested exercises, when they perform them

CONTACTS AND LOCATIONS:
Overall Officials: Karen Søgaard, PhD, Principal Investigator — University of Southern Denmark
Locations (2):
- Physical Activity and Health at Work, Department of Sports Science and Clinical Biomechanics, University of Southern Denmark, Odense, Denmark
- Norwegian University of Science and Technology, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mork PJ, Bach K; selfBACK Consortium. A Decision Support System to Enhance Self-Management of Low Back Pain: Protocol for the selfBACK Project. JMIR Res Protoc. 2018 Jul 20;7(7):e167. doi: 10.2196/resprot.9379. PMID 30030208
- [Derived] Kongstad LP, Overas CK, Skovsgaard CV, Sandal LF, Hartvigsen J, Sogaard K, Mork PJ, Stochkendahl MJ. Cost-effectiveness analysis of app-delivered self-management support (selfBACK) in addition to usual care for people with low back pain in Denmark. BMJ Open. 2024 Sep 5;14(9):e086800. doi: 10.1136/bmjopen-2024-086800. PMID 39242164
- [Derived] Bardal EM, Sandal LF, Nilsen TIL, Nicholl BI, Mork PJ, Sogaard K. Do age, gender, and education modify the effectiveness of app-delivered and tailored self-management support among adults with low back pain?-Secondary analysis of the selfBACK randomised controlled trial. PLOS Digit Health. 2023 Sep 22;2(9):e0000302. doi: 10.1371/journal.pdig.0000302. eCollection 2023 Sep. PMID 37738237
- [Derived] Svendsen MJ, Nicholl BI, Mair FS, Wood K, Rasmussen CDN, Stochkendahl MJ. One size does not fit all: Participants' experiences of the selfBACK app to support self-management of low back pain-a qualitative interview study. Chiropr Man Therap. 2022 Oct 3;30(1):41. doi: 10.1186/s12998-022-00452-2. PMID 36192724
- [Derived] Overas CK, Nilsen TIL, Nicholl BI, Rughani G, Wood K, Sogaard K, Mair FS, Hartvigsen J. Multimorbidity and co-occurring musculoskeletal pain do not modify the effect of the SELFBACK app on low back pain-related disability. BMC Med. 2022 Feb 8;20(1):53. doi: 10.1186/s12916-022-02237-z. PMID 35130898
- [Derived] Sandal LF, Bach K, Overas CK, Svendsen MJ, Dalager T, Stejnicher Drongstrup Jensen J, Kongsvold A, Nordstoga AL, Bardal EM, Ashikhmin I, Wood K, Rasmussen CDN, Stochkendahl MJ, Nicholl BI, Wiratunga N, Cooper K, Hartvigsen J, Kjaer P, Sjogaard G, Nilsen TIL, Mair FS, Sogaard K, Mork PJ. Effectiveness of App-Delivered, Tailored Self-management Support for Adults With Lower Back Pain-Related Disability: A selfBACK Randomized Clinical Trial. JAMA Intern Med. 2021 Oct 1;181(10):1288-1296. doi: 10.1001/jamainternmed.2021.4097. PMID 34338710
- [Derived] Rasmussen CDN, Svendsen MJ, Wood K, Nicholl BI, Mair FS, Sandal LF, Mork PJ, Sogaard K, Bach K, Stochkendahl MJ. App-Delivered Self-Management Intervention Trial selfBACK for People With Low Back Pain: Protocol for Implementation and Process Evaluation. JMIR Res Protoc. 2020 Oct 29;9(10):e20308. doi: 10.2196/20308. PMID 33118959
- [Derived] Sandal LF, Stochkendahl MJ, Svendsen MJ, Wood K, Overas CK, Nordstoga AL, Villumsen M, Rasmussen CDN, Nicholl B, Cooper K, Kjaer P, Mair FS, Sjogaard G, Nilsen TIL, Hartvigsen J, Bach K, Mork PJ, Sogaard K. An App-Delivered Self-Management Program for People With Low Back Pain: Protocol for the selfBACK Randomized Controlled Trial. JMIR Res Protoc. 2019 Dec 3;8(12):e14720. doi: 10.2196/14720. PMID 31793897
- See also: project webpage — http://www.selfback.eu

DOCUMENTS (2):
  • Study Protocol (2019-02-20): https://cdn.clinicaltrials.gov/large-docs/88/NCT03798288/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-08): https://cdn.clinicaltrials.gov/large-docs/88/NCT03798288/SAP_002.pdf